CLINICAL TRIAL: NCT05939674
Title: Effects of Flumazenil on Recovery After Total Intravenous Anesthesia With Remimazolam in Elderly Patients Undergoing Hip Joint Surgery: a Prospective Randomized Controlled Study.
Brief Title: Effects of Flumazenil on Recovery After Total Intravenous Anesthesia With Remimazolam
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, SANGWOOK SHIN, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 05-2023-134
Record Dates: First submitted 2023-06-22; First posted 2023-07-11 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Flumazenil Adverse Reaction; Remimazolam; Hip Joint; Elderly Patients
MeSH Terms: interventions — Flumazenil; Long-Term Synaptic Depression; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal saline group (Placebo Comparator): Participants are administered 3mL of 0.9% normal saline at the end of anesthesia
  Interventions: Drug: normal saline
- Flumazenil group (Active Comparator): Participants are administered 0.3mg(3mL) of flumazenil at the end of anesthesia
  Interventions: Drug: Flumazenil

INTERVENTIONS:
Drug: Flumazenil — During induction, patients will receive remimazolam 6mg/kg/h with remifentanil TCI 1~4 nanogram/mL. After patient loses consciousness, anesthesia will be maintained with remimazolam 1-2mg/kg/h combined with remifentanil. When procedure ends, infusion remimazolam stops and 0.3mg of flumazenil according to allocated groups.
  Other Names: Flumazenil, Flunil, Bukwang Pharm Co., Ltd
  Arms: Flumazenil group
Drug: normal saline — During induction, patients will receive remimazolam 6mg/kg/h with remifentanil TCI 1~4 nanogram/mL. After patient loses consciousness, anesthesia will be maintained with remimazolam 1-2mg/kg/h combined with remifentanil. When procedure ends, infusion remimazolam stops and 0.9% normal saline according to allocated groups.
  Other Names: Normal saline inj (JW)
  Arms: Normal saline group

SUMMARY:
Remimazolam is a medication that has the advantage of a short half-life and reversibility with flumazenil. In clinical situations, the use of flumazenil for the reversal of sedation is common, but there is no precise indication for its administration. In this study, we aim to investigate the necessity of routine flumazenil use after administering remimazolam for intravenous anesthesia.

DETAILED DESCRIPTION:
Remimazolam is a medication that has the advantage of a short half-life and reversibility with flumazenil.

Although there are advantages of using flumazenil, such as reduced recovery time and decreased occurrence of postoperative cognitive dysfunction (POCD), it can cause rebound sedation, ventricular arrhythmias, seizures, agitation, and gastrointestinal symptoms. Therefore, routine administration is not recommended.

However, in actual clinical situations, it is common to use flumazenil as a routine reversal agent for benzodiazepines, but there is no research on the routine use of flumazenil for reversing the effects of remimazolam in anesthesia or sedation.

Factors such as obesity, advanced age, and low plasma albumin concentration can prolong the time for extubation during anesthesia with remimazolam. Therefore, when considering the routine use of flumazenil in waking patients using remimazolam in elderly patients, these factors should be taken into account. However, there is also no specific indication for its accurate administration.

Therefore, this study aims to investigate the effects of flumazenil on recovery after total intravenous anesthesia with remimazolam in elderly patients undergoing hip joint surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years old scheduled for hip joint surgery

Exclusion Criteria:

* Patients with impaired consciousness or delirium before surgery
* Patients who are hemodynamically unstable before surgery
* Patients with a history of neurological or neuromuscular disorders or use of medications that affect neurological or neuromuscular function
* Patients who have taken sedatives (anti-anxiety medications, antipsychotics, antidepressants, sleep aids) within the past 24 hours
* Patients with known allergy to benzodiazepine, flumazenil
* Patients with galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Patients with hypersensitivity to Dextran40
* Patients who have been taking benzodiazepine for long term
* Patients with end stage renal disease requiring hemodialysis
* Patients with history of acute angle glaucoma
* Patients with alcohol or substance dependence
* ASA classification 4 or 5

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Difference in eye opening time between the two groups | Up to two hours
  Time, after stopping injection of remimazolam, to eye opening
Difference in extubation time between the two groups | Up to two hours
  Time, after stopping injection of remimazolam, to extubation

SECONDARY OUTCOMES:
Actual dose of flumazenil | Up to two hours, From end of anesthesia to discharge form the post-anestheic care unit
  Actual dose of flumazenil
Occurrence of re-sedation | Up to two hours, From end of anesthesia to discharge form the post-anestheic care unit
  Richmond Agitation Sedation Scale (RASS) score of -3 or lower(Score range: -5~+4, lower score means more sedated state)
Side effects of flumazenil usage | Up to two hours, From end of anesthesia to discharge form the post-anestheic care unit
  Number of Participants with Seizures, agitation, arrhythmias, gastrointestinal symptoms, post operative nausea and vomiting, and degree of pain

CONTACTS AND LOCATIONS:
Overall Officials: Sangwook Shin, MD. PhD, Study Director — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea